CLINICAL TRIAL: NCT06554600
Title: The Efficiency and Safety of Zanubrutinib in Combination With Polatuzumab Vedotin, Bendamustine and Rituximab in the Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma: a Prospective, Single-arm, Multicenter Study
Brief Title: A Study of Zanubrutinib in Combination With Polatuzumab Vedotin, Bendamustine and Rituximab in the Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2024279
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Refractory or Relapsed Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; polatuzumab vedotin; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pola-ZBR treatment (Experimental): Relapsed/refractory DLBCL were treated with 4 courses of Pola-ZBR regimen. Subjects achieving PR or CR were consolidated with autologous transplantation consolidation or the original regimen for 2 additional courses, and then given Zanubrutinib maintenance therapy for 1 year.
  Interventions: Drug: Zanubrutinib; Drug: Polatuzumab Vedotin; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — 160mg bid PO（d0-d20）
Drug: Polatuzumab Vedotin — Participants will receive a total of 4-6 cycles (a cycle being 21 days) of 1.8mg/kg Polatuzumab Vedotin on Day 2 of each cycle.
Drug: Bendamustine — Participants will receive a total of 4-6 cycles (a cycle being 21 days) of 70 mg/m2 Bendamustine on Days 2 and 3 of each cycle.
Drug: Rituximab — Participants will receive a total of 4-6 cycles (a cycle being 21 days) of 375 mg/m2 Rituximab on Day 1 of each cycle.

SUMMARY:
This is a prospective, multicenter, single-arm, open phase II study to explore the efficacy and safety of Zanubrutinib in combination with Polatuzumab Vedotin, bendamustine, and rituximab (Polo-ZBR) in subjects with relapsed/refractory diffuse large B-cell lymphoma. Subjects with relapsed/refractory DLBCL who met the inclusion/exclusion criteria were screened and treated with 4 courses of Pola-ZBR regimen after signing informed consent. Subjects achieving PR or CR were consolidated with autologous transplantation consolidation or the original regimen for 2 additional courses, and then given Zanubrutinib maintenance therapy for 1 year. The final follow-up was observed until 2 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 (inclusive);
* For patients with DLBCL confirmed by histopathology (which needs to be confirmed by specimens after this or past recurrence), the following DLBCL histology will be considered eligible for study enrollment:

DLBCL, NOS(includes GCB type and ABC type); T-cell rich large B-cell lymphoma; High-grade B-cell lymphoma with MYC and BCL-2 and/or BCL-6 rearrangement; High-grade B-cell lymphoma, NOS; Primary mediastinal (thymus) large B-cell lymphoma; EB virus positive DLBCL, NOS;HHV-8 positive DLBCL, NOS;

* Relapsed refractory patients, defined as those who had no response after first-line treatment (including immunochemotherapy, chemotherapy or hematopoietic stem cell transplantation) or relapsed or refractory after remission;
* There is at least one two-dimensional measurable lesion with a short diameter ≥1.0cm;
* Estimated survival time ≥3 months;
* The patient is informed and agrees to the program;
* ECOG score 0-2 points;
* Those who understand the procedure and content of the experiment, voluntarily participate in the study and sign the informed consent;
* Patients can follow up on schedule, communicate well with researchers and complete the trial according to the trial regulations;
* Confirm negative pregnancy test of female patients of childbearing age within 7 days before administration; Women and men in the reproductive period must agree to use medically recognized effective contraception throughout the treatment period and for 6 months after the end of the trial.

Exclusion Criteria:

* Active bleeding within 4 weeks prior to initial administration or anticoagulant therapy such as warfarin or vitamin K antagonists during the study period, or a tendency to bleed (such as esophageal varicose veins at risk of bleeding, locally active ulcerative lesions) or a clotting disorder deemed by the investigator;
* Surgical procedures have been performed within 6 weeks prior to the signing of the informed consent for the first dose of the trial drug, but tests for diagnostic purposes are not considered surgical procedures, and the insertion of a vascular access device will be exempt from this exclusion criteria;
* History of stroke and intracranial hemorrhage within 6 months before the first administration, except intracranial hemorrhage after surgery;
* Those who cannot stop or adjust moderate or strong CYP3A inhibitors;
* Have received organ transplantation or allogeneic stem cell transplantation;
* Previous or concurrent history of other malignant tumors;
* Chronic or currently active infectious diseases requiring systemic antibiotic, antifungal, or antiviral treatment (except EBV infections);
* Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, thrombotic diseases, connective tissue diseases and other diseases. Those who were not considered suitable for inclusion by the researchers;
* Laboratory test value at screening (unless due to lymphoma) : Leukocyte count < 3.5×109/L, neutrophils <1.5×109/L, platelets <80×109/L, hemoglobin <100g/L, ALT or AST were 2.5 times higher than the upper limit of normal, bilirubin was 1.5 times higher than the upper limit of normal, creatinine level was 1.5 times higher than the upper limit of normal;
* HbsAg positive patients need to check HBV-DNA < 104 to be enrolled. In addition, if HBsAg is negative but HBcAb is positive (regardless of HBsAb status), HBV-DNA testing is also required, and HBV-DNA results < 104 are required to be enrolled and continue treatment and monitoring of HBV-DNA. Patients with HCV antibody positive were required to check HCV-RNA quantitative DNA < 103 to be enrolled;
* HIV antibody, treponema pallidum antibody positive;
* Pregnant or lactating women;
* Those who have a history of drug use or drug abuse upon inquiry;
* Patient communication, understanding and cooperation are not enough, or compliance is poor, and it cannot be guaranteed that the program is carried out according to the requirements;
* Known allergy to the investigational drug or its related ingredients;
* Patients with past or current lymphoma central invasion;
* The patient is unable to swallow the capsule or has a disease or condition that severely affects gastrointestinal function, such as malabsorption syndrome, removal of the stomach or small intestine, or complete intestinal obstruction;
* Patients who could not stop using any other antitumor drugs within 2 weeks prior to medication in this study;
* Participants considered unsuitable for this clinical trial due to various other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate（ORR） | Up to 12 weeks
  The proportion of patients who achieved complete or partial response in efficacy evaluation at the end of induction treatment.

SECONDARY OUTCOMES:
Complete Response rate（CRR） | Up to 12 weeks
  The proportion of patients who achieved complete response in efficacy evaluation at the end of induction treatment.
Progression-free Survival（PFS） | Up to 2 years after enrollment
  PFS was defined as the period from date of enrollment until the date of disease progression, relapse, or death from any cause.
Overall Survival(OS) | Up to 2 years after enrollment
  OS was defined as the time from date of randomization until the date of death from any cause.
Percentage of Participants With Adverse Events (AEs) | Up to 12 weeks
  Toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No